CLINICAL TRIAL: NCT04921046
Title: Effect of Pretreatment of Lignocaine Versus Midazolam in the Prevention of Etomidate Induced Myoclonus
Brief Title: Effect of Pretreatment of Lignocaine Versus Midazolam in Prevention of Etomidate Induced Myoclonus.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, FIZZA BATOOL, Post graduate trainee Anesthesiology, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RMC Dissertation based article
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Myoclonic Jerk
MeSH Terms: conditions — Myoclonus | interventions — Lidocaine; Midazolam

STUDY DESIGN:
Intervention Model Description: two arm parallel assignment, two groups, receive two different drugs ;drug A and drug B to see the effect.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The test solutions were prepared in coded syringes and the observer was blinded to the groups as well as drugs .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Lignocaine (Active Comparator): Group of 112 patients ASA-I and II (American Society of Anesthesiology)ages from 25-44 undergoing elective surgical procedure.
  Interventions: Drug: lignocaine
- Group Midazolam (Active Comparator): Group of 112 patients ASA-I and II ages from 25-44 undergoing elective surgical procedure.
  Interventions: Drug: Midazolam 1 milligram Prefilled Syringe

INTERVENTIONS:
Drug: lignocaine — After giving lignocaine to a group of people, myoclonus was observed after the dose of etomidate given two minutes after lignocaine.
  Other Names: 2% lignocaine 1 ml
  Arms: Group Lignocaine
Drug: Midazolam 1 milligram Prefilled Syringe — after giving midazolam to the second group of people two minutes before etomidate dose, myoclonus was observed for one minute.
  Other Names: Dormicum
  Arms: Group Midazolam

SUMMARY:
This study is a randomized control trial and it was conducted to compare the effectiveness of pretreatment with lignocaine versus midazolam on the frequency of myoclonus associated with etomidate induction.

This was conducted in Holy Family Hospital Rawalpindi in a period of 6 months.

DETAILED DESCRIPTION:
INTRODUCTION:

General anaesthesia is loss of consciousness induced after administration of one or more general anaesthetic agent with overall aim of inducing sleep, amnesia, analgesia and skeletal muscles relaxation. Choosing an induction agent is a very vital step in commencing general anaesthesia1. Use of sedatives can prevent or minimize potentially harmful physiologic affects of airway manipulation that include increase in heart rate, BP, and raised intracranial pressure.

Etomidate, imidazole-derived, sedative-hypnotic agent, blocks neuroexcitation by its direct action on the gamma amino butyric acid (GABA) receptor complex1.Because of its many desirable properties like rapid onset of action, profound hypnosis, minimal histamine release, hemodynamic stability, minimal respiratory depression, and favorable cerebral effects, etomidate is considered as an ideal induction agent2. Concerns with etomidate include adrenal suppression and myoclonus3, 4.

30 to 60% of unpremedicated patients develop myoclonic movements after an induction dose (0.3 mg/kg) of etomidate1. Myoclonus is described as the involuntary contraction of some muscle fibers, leading to short observable movements of the body, more pronounced with the limbs5. In emergency scenarios, myoclonus can lead to increment in the chances of regurgitation and aspiration.

Various drugs like Lignocaine, Midazolam, Magnesium, Dezocine and dexmedetomidine have been used as pretreatment for reducing myoclonus after etomidate injection but the best drug for the purpose is yet to be discovered6, 7, 8, 9. Ideally a pretreatment drug should be short-acting, should affect respiration and hemodynamic minimally, and should not prolong the recovery period.

Lignocaine belongs to amide group of local anaesthetics.Lignocaine alters signal conduction in neuronal cell membrane8. Various studies have been conducted on lignocaine being used as a pretreatment drug; before propofol induction to reduce pain or etomidate to prevent myoclonus associated with etomidateinduction6.

Midazolam, a benzodiazepine, produce a calming effect on the brain and nerves 1, 10. Its various favorable effects include antiepileptic properties, anxiolysis, sedation, reduced attention and amnesia7. In a comparative study conducted by Singh KA (initials for first and second name of the author) et al, effect of pretreatment with lignocaine, midazolam and placebo were compared in prevention of etomidate induced myoclonus and the incidence was found to be 44%, 28% and 76% respectively5 (P<0.05). However, none of these studies have been conducted in Pakistan. The basic aim of my study is to compare the effectiveness of pretreatment with Lignocaine versus Midazolam on the frequency of myoclonus associated with etomidate induction, generate data regarding the effects, so that the more effective drug can be used routinely for the prevention of myoclonus associated with etomidate induction in routine.

METHODOLOGY:

After obtaining approval from the hospital ethics committee and written informed consent, 112 patient were recruited according to selection criteria in each group. All patients were assessed a day before surgery for anaesthesia fitness. Patient were prepared by fasting (8 h for solid foods, 4 hours for clear fluids).Patient were randomly divided into two equal groups by computer-generated numbers.

Group A received 1 ml of 2% lignocaine 2 min before induction with etomidate and Group B received 1 ml (1mg) of midazolam 2 min before induction with etomidate. On reaching the operating theater, standard monitoring were placed on all the participants, which included pulse oximeter, ECG and non-invasive blood pressure. A 20 G cannula with an intravenous line was maintained with 0.9% saline. Vitals such as pulse rate, blood pressure, respiratory rate, and oxygen saturation were recorded and taken as baseline readings. All patients were then preoxygenated with 100% oxygen for 3 min. Patients were divided randomly into two groups of 112 using computer generated random numbers. Group I received 1 ml of 2% lignocaine, and group II received 1 ml of midazolam (1 mg). The test solutions were prepared in coded syringes and were administered 2 min before etomidate induction (0.3 mg/kg) by an observer who was blinded to the allocation of the groups as well as the drug given to him. The time to the loss of eyelash reflex was recorded as the onset of induction, and an additional dose of etomidate was administered if necessary. The patients were observed continuously for myoclonic movements. The time of onset and the duration of myoclonus was observed. One minute post IV injection of etomidate and the observation of myoclonus, 0.5 mg/kg succinylcholine was administered to allow endotracheal tube placement. The vitals were observed after administration of test solution, after induction, and after endotracheal intubation every minute for five minutes, then every five minutes for fifteen minutes, and then every fifteen minutes till the surgery ends. Anesthesia was maintained with isoflurane (0.5-1%) and atracurium.

Data was collected on a standardized Proforma and analyze using SPSS-17 version (Statistical package for the social sciences). Mean ± SD (standard deviation) was calculated for quantitative variables lik age, weight and BMI. Qualitative variables like gender, myoclonus wer expressed as frequencies and percentages. Chi-square was used to compare th frequency of myoclonus in two groups. A P value less than 0.05 was consider statistically significant. Effect modifiers like age and gender were controlled b stratification. Post-stratification Chi-square test was applied.

ELIGIBILITY:
Inclusion Criteria:

* ASA-I / ASA-II
* any gender >20-45 years
* undergoing elective surgical procedure.

Exclusion Criteria:

* Patient who refused
* those with any neurological or psychiatric disorders
* morbid obesity
* drug allergies
* pregnant patients

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Occurrence and Frequency of Myoclonus | Immediately after giving etomidate dose.
  involuntary contracting muscle fibers leading to short observable movements more pronounced with the limbs measured by observation by an observer.
Occurrence and Frequency of Myoclonus | 20 seconds after giving etomidate dose.
  involuntary contracting muscle fibers leading to short observable movements more pronounced with the limbs measured by observation by an observer.
Occurrence and Frequency of Myoclonus | 40 seonds after giving etomidate dose.
  involuntary contracting muscle fibers leading to short observable movements more pronounced with the limbs measured by observation by an observer.
Occurrence and Frequency of Myoclonus | 60 seconds after giving etomidate dose.
  involuntary contracting muscle fibers leading to short observable movements more pronounced with the limbs measured by observation by an observer.

CONTACTS AND LOCATIONS:
Overall Officials: Fizza Batool, FCPS, Principal Investigator — Rawalpindi Medical College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devlin RJ, Kalil D. Etomidate as an Induction Agent in Sepsis. Crit Care Nurs Clin North Am. 2018 Sep;30(3):e1-e9. doi: 10.1016/j.cnc.2018.05.004. Epub 2018 Jul 13. PMID 30286947
- [Background] Malapero RJ, Zaccagnino MP, Brovman EY, Kaye AD, Urman RD. Etomidate derivatives: Novel pharmaceutical agents in anesthesia. J Anaesthesiol Clin Pharmacol. 2017 Oct-Dec;33(4):429-431. doi: 10.4103/0970-9185.222521. PMID 29416230
- [Background] Du X, Zhou C, Pan L, Li C. Effect of dexmedetomidine in preventing etomidate-induced myoclonus: a meta-analysis. Drug Des Devel Ther. 2017 Feb 8;11:365-370. doi: 10.2147/DDDT.S121979. eCollection 2017. PMID 28223779
- [Background] Forman SA. Clinical and molecular pharmacology of etomidate. Anesthesiology. 2011 Mar;114(3):695-707. doi: 10.1097/ALN.0b013e3181ff72b5. PMID 21263301
- [Background] Apartis E, Vercueil L. To jerk or not to jerk: A clinical pathophysiology of myoclonus. Rev Neurol (Paris). 2016 Aug-Sep;172(8-9):465-476. doi: 10.1016/j.neurol.2016.07.013. Epub 2016 Aug 24. PMID 27568397
- [Background] Lang B, Zhang L, Li F, Lin Y, Zhang W, Yang C. Comparison of the efficacy and safety of remifentanil versus different pharmacological approaches on prevention of etomidate-induced myoclonus: a meta-analysis of randomized controlled trials. Drug Des Devel Ther. 2019 May 9;13:1593-1607. doi: 10.2147/DDDT.S200200. eCollection 2019. PMID 31190739
- [Background] Gupta P, Gupta M. Comparison of different doses of intravenous lignocaine on etomidate-induced myoclonus: A prospective randomised and placebo-controlled study. Indian J Anaesth. 2018 Feb;62(2):121-126. doi: 10.4103/ija.IJA_563_17. PMID 29491517
- [Background] Sedighinejad A, Naderi Nabi B, Haghighi M, Biazar G, Imantalab V, Rimaz S, Zaridoost Z. Comparison of the Effects of Low-Dose Midazolam, Magnesium Sulfate, Remifentanil and Low-Dose Etomidate on Prevention of Etomidate-Induced Myoclonus in Orthopedic Surgeries. Anesth Pain Med. 2016 Apr 2;6(2):e35333. doi: 10.5812/aapm.35333. eCollection 2016 Apr. PMID 27247915
- [Background] Niedermirtl F, Eberhardt M, Namer B, Leffler A, Nau C, Reeh PW, Kistner K. Etomidate and propylene glycol activate nociceptive TRP ion channels. Mol Pain. 2018 Jan-Dec;14:1744806918811699. doi: 10.1177/1744806918811699. Epub 2018 Oct 22. PMID 30345869
- [Background] Wu GN, Xu HJ, Liu FF, Wu X, Zhou H. Low-Dose Ketamine Pretreatment Reduces the Incidence and Severity of Myoclonus Induced by Etomidate: A Randomized, Double-Blinded, Controlled Clinical Trial. Medicine (Baltimore). 2016 Feb;95(6):e2701. doi: 10.1097/MD.0000000000002701. PMID 26871805
- [Background] Safavi M, Honarmand A, Sahaf AS, Sahaf SM, Attari M, Payandeh M, Iazdani A, Norian N. Magnesium sulfate versus Lidocaine pretreatment for prevention of pain on etomidate injection: A randomized, double-blinded placebo controlled trial. J Res Pharm Pract. 2015 Jan-Mar;4(1):4-8. doi: 10.4103/2279-042X.150044. PMID 25710044
- [Background] Huter L, Schreiber T, Gugel M, Schwarzkopf K. Low-dose intravenous midazolam reduces etomidate-induced myoclonus: a prospective, randomized study in patients undergoing elective cardioversion. Anesth Analg. 2007 Nov;105(5):1298-302, table of contents. doi: 10.1213/01.ane.0000287248.25610.c0. PMID 17959958
- [Background] Ye Young Yang, Sae Jin Choi, Hae Ja Kim, Soo Chang Son. The effect of midazolam, fentanyl and a small dose of etomidate for prevention of myoclonus during induction of anesthesia with etomidate. Clinical Research Article. Korean J Anesthesiol. 2000;39(2):1-66-171
- [Result] Singh Ka, Ruchi G, Singh KA, Kaur BT Efficacy of lignocaine versus midazolam in controlling etomidate-induced myoclonus: a randomized placebo-controlled study. Ai Shams Med J 2014;7(3):460-4
- [Result] Lang B, Zhang L, Yang C, Lin Y, Zhang W, Li F. Pretreatment with lidocaine reduces both incidence and severity of etomidate-induced myoclonus: a meta-analysis of randomized controlled trials. Drug Des Devel Ther. 2018 Oct 4;12:3311-3319. doi: 10.2147/DDDT.S174057. eCollection 2018. PMID 30323563
- [Result] Schwarzkopf KR, Hueter L, Simon M, Fritz HG. Midazolam pretreatment reduces etomidate-induced myoclonic movements. Anaesth Intensive Care. 2003 Feb;31(1):18-20. doi: 10.1177/0310057X0303100103. PMID 12635389